CLINICAL TRIAL: NCT02999607
Title: Brain Glucose Metabolism in Healthy Subjects and Depressive Patients During Transcranial Direct Current Stimulation
Brief Title: Brain Glucose Metabolism During Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc. Prof. Priv.-Doz., Medical University of Vienna
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 3.0.30.11.16
Record Dates: First submitted 2016-12-18; First posted 2016-12-21 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Depression
Keywords: Transcranial direct current stimulation; Positron emission tomography
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- active transcranial direct current stimulation (Experimental): Stimulation at three different intensities during FDG-PET scan
  Interventions: Other: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Comparator to active arm
  Interventions: Other: transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — 0.5 mA, 1mA, 2mA for 10 minutes each

SUMMARY:
With this study we will be able to dose-dependently measure real-time glucose metabolism changes after non-invasively stimulating superficial parts of the dlPFC, a commonly used target in therapeutic tDCS applications. This will provide further insight if and how tDCS is capable to change one of most reliable parameters of brain metabolism.

DETAILED DESCRIPTION:
With this study, we will be able to substantiate if regional and whole brain glucose metabolism is affected by tDCS, assess the amount of signal change in relation to different currents and measure differences in glucose metabolism under stimulation reactivity between healthy subjects and depressive patients. The objective is to investigate the changes of regional cerebral metabolic rate of glucose (rCMRglu) in the brain after transcranial direct current stimulation in healthy subjects and depressive patients. The design is a cross-sectional proof of principle study in 20 healthy subjects and 20 depressed patients. During the PET scan tDCS will be applied with varying stimulus intensity. Furthermore, subjects will undergo a second PET scan with single-blind sham stimulation in order to validate the effects of tDCS. rCMRglu will be quantified using voxel-wise and ROI-based approaches. Changes in rCMRglu associated with tDCS-application will be calculated with a general linear model in a ramp function of the task-specific glucose uptake, according to previous work in our group. Exploratory statistical testing will be done using a paired samples t-test between task and rest conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

- Aged 18 to 55 years Somatic and psychiatric health based on medical history, physical examination, ECG, laboratory screening, SCID-I and II Willingness and competence to complete the informed consent process

Depressed Patients:

Current major depressive episode during unipolar major depression (MD) according to SCID-I (with HAMD>17) No other concomitant axis-I disease apart from anxiety disorder, which must be secondary to MD Standard antidepressant medication stable during the last 4 weeks

Exclusion Criteria:

* Concomitant major medical or neurological illness, including history of seizures Any current substance abuse disorder according to DSM-V (urinary test and history) including current sedative usage in MDD patients ECT, TMS or NMDA-antagonists (ketamine) during the past 6 months. Current augmentation with anti-epileptics, or other drugs affecting seizure threshold Failure to comply with the study protocol or follow the instructions of the investigators Pregnancy Participants with previous total radiation exposure dose of 30mSv over the last 10 years (according to legislation on radiation protection).

Left-handedness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
FDG-rCMRglu | 70 minutes
  regional cerebral metabolic rate of glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria